CLINICAL TRIAL: NCT01019915
Title: Effect of Cardiac Resynchronization Therapy on Skeletal Muscle Histology, Neuroendocrine Activation and Inflammatory Response
Brief Title: Effect of Cardiac Resynchronization Therapy (CRT) on Skeletal Muscle Histology, Neuroendocrine Activation and Inflammatory Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University of Tromso (Other); University of Oslo (Other); The Royal Norwegian Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRT-AIL-SUS 2009
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2011-06

CONDITIONS: Skeletal Muscle Changes After Crt
Keywords: CRT; heart failure; left bundle branch block; skeletal muscle; cytokines; VO2; pgc1alpha
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heart failure patients. Intervention CRT (Other): CRT implantation in heart failure. Effect of intervention after 6 months of treatment.
  Interventions: Device: CRT

INTERVENTIONS:
Device: CRT — Insertion of CRT in patients with left bundle branch block. Assessment of skeletal muscle and infalmmatory profile

SUMMARY:
Heart failure patients with left bundle branch block have a poor prognosis. Biventricular pacing which synchronize the heart pump action is associated with improved functional capacity. This study aims to evaluate the basic changes in skeletal muscle functioning after a period of biventricular pacing in 21 patients with heart failure.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is the most common hospital discharge diagnosis in elderly patients . Fatigue and dyspnea with exercise intolerance and a poor quality of life are the main characteristics of this syndrome , and it is associated with substantial mortality and morbidity , .

Although the systolic dysfunction has been recognized as the primum movens of CHF, it is now generally accepted that the progression of the syndrome is not solely related to the pump failure.

The neuro-endocrine model has reached a wide consensus as one of the basic mechanisms for progressive heart failure based on the good results obtained by ACE-inhibitor therapy . A decade ago the cytokine model was added to explain the syndrome of heart failure . The cytokines are highly potent endogenous peptides produced by different cell types . Elevated levels might be markers for cardiac cachexia, but they may also play an important role in the mechanism of CHF progression . Subsequently, the muscle hypothesis was proposed as an explanation for the deconditioning in CHF patients . In skeletal muscle from healthy individuals there is a balanced distribution between type I fibres (aerobic), type IIA fibres (both aerobic and anaerobic) and type IIB fibres (mostly anaerobic). In CHF a shift to type II fibres and a reduced capillary density as well as a reduced cytochrome oxidase activity is observed, but the mechanisms leading to such a shift have not been clarified . Deconditioning may be an important factor aggravating the underlying pathophysiology in CHF and exercise training has been shown to improve exercise performance and to reduce symptoms in this population . This is partly mediated by activation of the Protein PGC-1, a critical factor coordinating the activation of metabolic genes required for substrate utilization and mitochondrial biogenesis . The increase in this enzyme has been highly correlated to increase in peak VO2 after a aerobic interval training program in heart failure .

One would expect that an improvement in exercise performance following improvement in central hemodynamics with cardiac resynchronization therapy (CRT) would be associated with improved muscular blood flow and energy metabolism. However, so far no reports have been published on the skeletal muscle response to CRT. The purpose of this study was to evaluate the effect of 6 months CRT pacing on skeletal muscle histology and mitochondrial mass and the association of these changes to alterations in functional capacity as measured with peak VO2. Moreover, we also sought to assess the relationship between changes in skeletal muscle and alterations in the inflammatory response in serum and in skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure, left bundle branch block

Exclusion Criteria:

* serious comorbidity including systemic inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
capillary density | finnished
  To assess if CRT improves skeletal muscle cappillary density

CONTACTS AND LOCATIONS:
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Derived] Larsen AI, Valborgland T, Ogne C, Lindal S, Halvorsen B, Munk PS, Kvaloy JT, Aukrust P, Yndestad A. Plasma tumour necrosis factor correlates with mRNA expression of tumour necrosis factor and mitochondrial transcription factors in skeletal muscle in patients with chronic heart failure treated with cardiac resynchronization therapy: potential role in myopathy. Eur J Prev Cardiol. 2020 Dec;27(19):2362-2366. doi: 10.1177/2047487319855796. Epub 2019 Jun 8. No abstract available. PMID 31389718
- [Derived] Larsen AI, Lindal S, Myreng K, Ogne C, Kvaloy JT, Munk PS, Aukrust P, Yndestad A, Dickstein K, Nilsen DW. Cardiac resynchronization therapy improves minute ventilation/carbon dioxide production slope and skeletal muscle capillary density without reversal of skeletal muscle pathology or inflammation. Europace. 2013 Jun;15(6):857-64. doi: 10.1093/europace/eus428. Epub 2013 Jan 15. PMID 23322010